CLINICAL TRIAL: NCT00298766
Title: An Open-Label Phase 1/2 Study of VELCADE for Injection in Subjects With Light-Chain (AL)-Amyloidosis
Brief Title: Open-Label Phase 1/2 Study of VELCADE for Injection in Patients With Light-chain (AL)-Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-CAN-2007
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Results first posted 2010-08-13 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Bortezomib

ARMS (1):
- 1 (Experimental): VELCADE
  Interventions: Drug: VELCADE

INTERVENTIONS:
Drug: VELCADE — Once weekly at: 0.7, 1.0, 1.3 or 1.6 mg/m2
  Or
  Twice-weekly at: 0.7, 1.0, or 1.3 mg/m2
  Other Names: Bortezomib

SUMMARY:
This is a phase 1/2 open-label, dose-escalation study investigating single-agent therapy with VELCADE in patients with previously treated systemic AL-amyloidosis who require further treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 18 y/o and older
2. Female patients must be practicing an effective method of birth control
3. Biopsy-proven AL-amyloidosis
4. Must have been previously treated (failed at least 1 previous treatment) and in the opinion of the physician, patient requires further treatment

Exclusion Criteria:

1. Hypersensitivity to boron or mannitol
2. Prior treatment with VELCADE
3. Patient requires other concomitant chemotherapy, radiotherapy or ancillary therapy considered investigational
4. Uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-06; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Winship Cancer Center - Emory Clinic School of Medicine, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - MSKCC, New York, New York

REFERENCES:
- [Derived] Reece DE, Hegenbart U, Sanchorawala V, Merlini G, Palladini G, Blade J, Fermand JP, Hassoun H, Heffner L, Kukreti V, Vescio RA, Pei L, Enny C, Esseltine DL, van de Velde H, Cakana A, Comenzo RL. Long-term follow-up from a phase 1/2 study of single-agent bortezomib in relapsed systemic AL amyloidosis. Blood. 2014 Oct 16;124(16):2498-506. doi: 10.1182/blood-2014-04-568329. Epub 2014 Sep 8. PMID 25202139
- [Derived] Reece DE, Hegenbart U, Sanchorawala V, Merlini G, Palladini G, Blade J, Fermand JP, Hassoun H, Heffner L, Vescio RA, Liu K, Enny C, Esseltine DL, van de Velde H, Cakana A, Comenzo RL. Efficacy and safety of once-weekly and twice-weekly bortezomib in patients with relapsed systemic AL amyloidosis: results of a phase 1/2 study. Blood. 2011 Jul 28;118(4):865-73. doi: 10.1182/blood-2011-02-334227. Epub 2011 May 11. PMID 21562045
- [Derived] Reece DE, Sanchorawala V, Hegenbart U, Merlini G, Palladini G, Fermand JP, Vescio RA, Liu X, Elsayed YA, Cakana A, Comenzo RL; VELCADE CAN2007 Study Group. Weekly and twice-weekly bortezomib in patients with systemic AL amyloidosis: results of a phase 1 dose-escalation study. Blood. 2009 Aug 20;114(8):1489-97. doi: 10.1182/blood-2009-02-203398. Epub 2009 Jun 4. PMID 19498019

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Agent VELCADE: Bortezomib 0.7, 1.0, 1.3 and 1.6 mg/m^2 once weekly (QW) 4 doses in a 5 week cycle, and 0.7, 1.0, 1.3 mg/m^2 twice weekly (BIW) 4 doses in a 3 week cycle
Period: Overall Study
Arm/Group | Single Agent VELCADE
Started | 70
Completed | 24
Not Completed | 46
Not completed — Adverse Event | 18
Not completed — Death | 2
Not completed — Withdrawal by Subject | 9
Not completed — Treatment ongoing | 4
Not completed — Progression of amyloid markers | 4
Not completed — Deterioration in KPS and organ function | 1
Not completed — Subjects overall condition deterioration | 4
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 35
  Canada | 8
  France | 3
  Germany | 11
  Italy | 9
  Spain | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Maximum Tolerated Dose (MTD) was defined as the highest dose level that has 0/1 out of 6 patients experiences Dose Limited Toxicity (DLT). MTD is defined separately for QW and BIQ dose cohorts.
  DLT was defined as adverse events occurring during Cycle 1 and: (1) related to VELCADE, (2) Grade 4 thrombocytopenia or neutropenia, (3) Grade 3 or higher nonhematologic toxicity.
Time Frame: 5 weeks in once weekly (QW) dose cohorts and 3 weeks in twice weekly (BIW) dose cohorts
Population: Phase 1 Safety Population includes all subjects who received at least one dose of VELCADE in phase 1 dose escalation cohorts
Measure: Number; unit: participants with DLT
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 31
participants with DLT | 2

2. Primary Outcome: Subjects With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events observed during outcome measure time frame
Time Frame: from first study-related procedure to 30 days after last dose of study medication
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 70
participants | 70

3. Secondary Outcome: Best Confirmed Hematologic Responders
Description: Hematologic response was determined by the investigator per the response criteria for immunoglobulin light chain amyloidosis by Gertz (2005). It include Complete and Partial Responders (CR+PR). CR requires serum and urine negative for a monoclonal protein by immunofixation and free light chain ratio normal. PR requires: 1. reduction in quantitative serum M-protein by 50% if baseline value is at least 0.5 g/dL, 2. if light chain is detected in the urine (with a consistent peak and >100 mg/ 24 hours), then 50% reduction is required, 3. if free light chain >10 mg/dL, reduction by 50% is required.
Time Frame: from first dose of study medication to end of study visit
Population: Efficacy population included all treated subjects with an evaluable post baseline resposne assessment in the MTD cohorts (1.6 mg/m^2 QW and 1.3 mg/m^2 BIW).
Measure: Number; unit: participants responded
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 49
participants responded | 33

4. Primary Outcome: Subjects With Serious Treatment Emergent Adverse Events
Description: Serious treatment emergent adverse events observed during outcome measure time frame
Time Frame: from first study-related procedure to 30 days after last dose of study medication
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 70
participants | 25

5. Primary Outcome: Subjects Grade 3/4/5 Treatment Emergent Adverse Events
Description: Grade 3/4/5 treatment emergent adverse events observed during outcome measure time frame.
  Grade is determined according to Common Terminology Criteria for Adverse Event (CTCAE) Version 3.0.
Time Frame: from first study-related procedure to 30 days after last dose of study medication
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 70
participants | 43

6. Primary Outcome: Subjects With Treatment Emergent Adverse Events Leading to Treatment Termination
Description: Treatment emergent adverse events observed during outcome measure time frame leading to treatment termination
Time Frame: from first study-related procedure to 30 days after last dose of study medication
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Single Agent VELCADE
Number analyzed (Participants) | 70
participants | 23

ADVERSE EVENTS:
Time Frame: from first study-related procedure to 30 days after last dose of study medication
Arm/Group | Single Agent VELCADE
Serious Adverse Events (participants affected / at risk) | 25/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent VELCADE (N=70)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure cogestive (Cardiac disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Autonomic neuropathy (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Penal impairment (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent VELCADE (N=70)
Anaemia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 4
Palpitations (Cardiac disorders) | 5
Conjunctival haemorrhage (Eye disorders) | 5
Conjunctivitis (Eye disorders) | 6
Dry eye (Eye disorders) | 4
Vision blurred (Eye disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 9
Chest pain (General disorders) | 4
Chills (General disorders) | 7
Early satiety (General disorders) | 4
Influenza like illness (General disorders) | 5
Oedema (General disorders) | 15
Oedema peripheral (General disorders) | 16
Pain (General disorders) | 4
Pyrexia (General disorders) | 12
Bronchitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 5
Periorbital haematoma (Injury, poisoning and procedural complications) | 4
Anorexia (Metabolism and nutrition disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 16
Hypoaesthesia (Nervous system disorders) | 7
Neuropathy peripheral (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 17
Peripheral sensory neuropathy (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 5
Night sweats (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 4
Phlebitis (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No